CLINICAL TRIAL: NCT05157607
Title: Family Connections for Caregivers of People With Suicidal Behavior: Study Protocol of a Randomized Control Trial.
Brief Title: Family Connections for Caregivers of People With Suicidal Behavior
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Valencia (Other)
Collaborators: Universitat Jaume I (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UV-1623849
Record Dates: First submitted 2021-12-01; First posted 2021-12-15 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Relatives
Keywords: Family Connections; Suicidal Behavior Disorder; Suicide Attempts; Caregivers; Dialectical Behavior Therapy
MeSH Terms: conditions — Suicide, Attempted | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized Control Trial, efficacy Study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Family Connections Protocol for Relatives of Patients with SBD. (Experimental): The intervention lasts three months and includes 12 sessions with a weekly two-hour group format. The FC program is divided into six modules:
  Module 1: Up-to-date information and research on suicide (Epidemiology, frequency, Risk factors, protective factors).
  Module 2: Psychoeducation on the development of suicide, explanatory theories, available treatments, comorbidity.
  Module 3: Emotional regulation skills, skills of acceptance, validation, approach, awareness, and to decrease emotional reactivity.
  Module 4: Skills to improve the quality of relationships in family interactions (letting go of guilt and anger, acceptance skills in relationships).
  Module 5: Communication skills and effective self-expression. Module 6: Problem management and making safe plans for crisis management.
  Interventions: Behavioral: Family Connections Protocol for Relatives of Patients with SBD.
- Treatment as Usual Optimized Protocol (TAU-O). (Active Comparator): Family members in this condition will continue to receive their treatment as usual in their care center of reference. In addition, we will optimize the treatment based on the recommendations of the international guidelines for the treatment of suicide. There will be one three-hour session in group format with the following component:
  Module 1: Updated information and research on suicide (Epidemiology, frequency, Risk factors, protective factors). Psychoeducation on the development of Suicide, Explanatory theories. Available treatments, and comorbidity.
  Interventions: Behavioral: Treatment as Usual Optimized Protocol (TAU-O)

INTERVENTIONS:
Behavioral: Family Connections Protocol for Relatives of Patients with SBD. — Family Connections is a Dialectical Behavioral Therapy. All the modules include practice exercises, video viewing, and homework assignments. In addition, throughout the program, with the aim of increasing social support, the FC-SBD program provides a forum where participants can stay in touch and share common problems and solutions.
  Arms: Family Connections Protocol for Relatives of Patients with SBD.
Behavioral: Treatment as Usual Optimized Protocol (TAU-O) — Participants will receive the usual treatment in their mental health service and will also receive a psychoeducation session of approximately 3 hours where the predictive and protective factors of suicidal behavior will be explained.
  Arms: Treatment as Usual Optimized Protocol (TAU-O).

SUMMARY:
The aim of our study is to verify the efficacy of the Family Connections intervention for relatives of people diagnosed with suicidal behavior disorder in a randomized control trial with a Spanish participants.

DETAILED DESCRIPTION:
Family members of people who have attempted suicide feel guilty, afraid, hopeless, depression and anxiety. The needs of family members of people with suicide attempts are not adequately addressed in the current treatments for people with suicide attempts. Therefore, it is necessary to help the relatives of people with suicidal behaviors to reduce the discomfort and burden they experience by giving them information and skills to improve their relationship with patients. Family Connections (FC) is a program that has been shown to be effective in reducing burden, depression, and anxiety, and in increasing dominance and validating behaviors in relatives of people with borderline personality disorder. However, there are no Randomized Control Trials that demonstrate the efficacy of FC program in patients with suicide attempts. In a previous study, FC was adapted in an open trial with relatives of people who had attempted suicide. The results of this pilot study suggest that the FC program tailored to relatives of patients with suicide attempts may be effective in improving well-being and reducing the burden of illness in relatives.

Our research team adapted FC for relatives of people diagnosed with suicidal behavior disorder (SBD) for delivery in the Spanish population. The FC-SCD program contains 12 two-hour sessions held once a week. The first aim is to verify the efficacy of the FC intervention for relatives of people diagnosed with SBD in a randomized control trial with a Spanish sample of participants from mental health services. The second objective is to analyze the feasibility and acceptance of FC-SBD in relatives. The third aim is to analyze whether the changes produced in the psychological variables in the relatives after the intervention are related to changes in the psychological variables of the patients. This paper presents the study protocol. The study design consists of a two-arm randomized controlled trial, there will be two conditions: Family Connections (FC-SBD) or Treatment as usual optimized (TAU-O). Participants will be relatives of patients who meet DSM-5 criteria for SBD. The caregivers' primary outcome measures will be the BAS. Secondary outcomes will be DASS-21, FES, DERS, QoL. The patient's primary outcome measures will be the INQ, PHQ-9, OASIS, VIRS, LUMP. Participants will be assessed at pretreatment, post-treatment, and 6-month follow-up. The intention-to-treat principle will be used when analyzing data, using mixed-effects models with full information and maximum likelihood estimation.

ELIGIBILITY:
Inclusion Criteria:

* Being a caregiver of one patient with a diagnosis of Suicide Behavior Disorder
* Understand spoken and written Spanish;
* Signing the informed consent.

Exclusion Criteria:

* The presence of a diagnosis of severe mental disorder in the caregivers as: Psychosis, schizophrenia, substance dependence, or high suicide ideation.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
Burden assessment scale (BAS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  This 19-item scale assesses two dimensions of caregiver burden of a loved one's illness (objective and subjective) in the past six months. The items are rated on a 4-point Likert scale (1-4), where higher scores indicate higher levels of illness burden. The psychometric properties of this scale are adequate, with an internal reliability between .89 and .91 and adequate validity.

SECONDARY OUTCOMES:
Family empowerment scale (FES) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  This scale has a total of 34 items. It is composed of three subscales referring to attitudes, knowledge, and behaviors related to (1) Family, (2) the Service System, and (3) Community Participation. The items are rated on a Likert scale (1-5), where higher scores show greater feelings of empowerment. Both the validity and reliability of this scale are adequate, and the internal consistency of the subscales shows coefficients between α = .87 and α =.88.
Depression, anxiety, and stress scale (DASS-21) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  We have used the short, validated Spanish version with 21 items on the frequency of negative emotional symptoms in the past week. The items are rated on a Likert scale (0-3) where the higher the score, the higher the frequency of symptoms of depression, anxiety, and/or stress. The internal consistency of the scale was excellent, with Cronbach's alphas for the DASS-21 subscales: Depression (α = .94), Anxiety (α = .87) and Stress (α = .91)
Difficulties in emotion regulation scale - Spanish version | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  We used the Spanish validation containing 28 items. This questionnaire is divided into five subscales: (1) Lack of emotional control, (2) Life interference, (3) Emotional inattention, (4) Emotional confusion, and (5) Emotional rejection. The items are rated on a Likert scale (1-5) where higher scores indicate greater difficulty in regulating emotions. Psychometric properties are excellent, with an internal consistency of α = .93 and test-retest reliability of pl = .74, p < .001
Quality of life index-Spanish version (QLI-Sp) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  It consists of a 10-item index of perceived quality of life. It refers to physical and emotional well-being, functioning at work, satisfaction with personal relationships and self-independence, support in the community and from an emotional point of view, spiritual well-being, and perceived overall quality of life. The items are rated on a Likert scale (0-10) where higher scores indicate higher perceived quality of life. The psychometric properties are good for both internal consistency (α = .89) and test-retest reliability (r = 0.87).
Opinion and Expectations of Treatment Scale (OTSM) | Changes will be assessed from pre-treatment to immediately after the intervention
  This scale was designed and developed by members of the research team and constructed from an adaptation of another opinion and expectations questionnaire [49]. The constructs this scale assesses are: opinion, acceptance and satisfaction with the skills training program, and the changes in the participants after the completion of each module. The questions refer to the rationale for the intervention, recommendation of the program, satisfaction with the program, usefulness and expectations of the skills training. The items are rated on a Likert-type scale ranging from 0 "Not at all" to 10 "Very much".
Register of critical incidents with the family member with SBD | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  his register was developed ad hoc for this study. The questions recorded are the following: frequency of suicide attempts in the past six months, number of days of self-harm in the past six months, number of episodes of verbal/physical violence with caregivers in the past six months; frequency of visits to the psychiatric emergency room in the past six months, frequency of therapy sessions conducted out of schedule in the past six months (face-to-face, phone calls, etc.).

OTHER OUTCOMES:
Register of critical incidents with the patient member with SBD | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  This register was developed ad hoc for this study. The questions recorded are the following: frequency of suicide attempts in the past six months, number of days of self-harm in the past six months, number of episodes of verbal/physical violence with caregivers in the past six months; frequency of visits to the psychiatric emergency room in the past six months, frequency of therapy sessions conducted out of schedule in the past six months (face-to-face, phone calls, etc.).
Interpersonal Needs Questionnaire (INQ) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  We use the Spanish version of this 15-item questionnaire that assesses the degree of dissatisfaction with their need to belong (frustrated belonging) and the degree to which they perceive themselves as a burden to others (perceived burden). The items are rated on a Likert-type scale (1-7) where higher scores indicate higher levels of frustrated belonging and perceived burden to others. Psychometric properties were good: scale reliability was very good (perceived burden, α = 0.96; and frustrated belonging, α = 0.78).
Patient Health Questionnaire (PHQ-9) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  It consists of a nine-item questionnaire that assesses depressive symptoms in the past two weeks. Specifically, it includes the DSM-IV diagnostic criteria A for major depressive disorder (American Psychiatric Association, 2000). The items are rated on a Likert scale (0-3) where higher scores indicate higher frequency of depressive symptoms. The severity of depression on this questionnaire is measured through the total score, which can be categorized as none or minimal, mild, moderate, moderately severe, and severe. Validity has been adequate, with a sensitivity of 88% and a speciﬁcity of 88% for major depression
Overall Anxiety Severity and Impairment Scale (OASIS | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  We use the Spanish version of this questionnaire, which consists of a five-item instrument that assesses the frequency and intensity of anxiety symptoms in the past week. In addition, it measures interference in work and academic, social, and daily life domains, as well as avoidance behaviors. The items are rated on a Likert-type scale (0-4). The psychometric properties are good in terms of internal consistency (α= 0.86), convergent and discriminant validity, and sensitivity to change (α= 0.86).
Validating and Invalidating Responses Scale (VIRS) | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  It consists of a 16-item scale on the validation and invalidation of family members' responses about their loved ones. It is divided into two subscales (validation and invalidation), and the items are rated on a Likert scale (0-4) where higher scores indicate higher perceived validation or higher perceived invalidation (depending on the subscale).
Lum Emotional Availability of Parents | Changes will be assessed from pre-treatment to immediately after the intervention, and also at 6-month follow-up.
  This 15-item questionnaire measures the perceived emotional availability of primary caregivers. The items are rated on a Likert scale (1-6) where higher scores indicate greater emotional availability of caregivers. Psychometric properties were excellent for both subscales (mother, α = .9; and father, α = .93). In addition, test-retest reliability was also adequate for the mother's subscale (r = .92) and the father's subscale (r = .85).

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Fernández Felipe, PhDStudent, Principal Investigator — Universitat Jaume I; Sara Fonseca, PhDStudent, Principal Investigator — University of Valencia; Azucena Garcia-Palacios, PhD, Principal Investigator — Universitat Jaume I; Sandra Perez, PhD, Principal Investigator — Universitat de Valencia; Rosa Baños, PhD, Principal Investigator — Universitat de Valencia; Cristina Botella Arbona, PhD, Principal Investigator — Universitat Jaume I; Joaquin Garcia-Alandete, PhD, Principal Investigator — Universitat de Valencia
Locations (1):
- University of Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will be available after deidentification
Supporting Information: Study Protocol, SAP, CSR
Time Frame: The data will be available immediately following publication
Access Criteria: The data will be available to anyone who wishes to access them.

REFERENCES:
- [Background] Hoffman PD, Fruzzetti AE. Advances in interventions for families with a relative with a personality disorder diagnosis. Curr Psychiatry Rep. 2007 Feb;9(1):68-73. doi: 10.1007/s11920-007-0012-z. PMID 17257517
- [Background] Hoffman PD, Fruzzetti AE, Buteau E, Neiditch ER, Penney D, Bruce ML, Hellman F, Struening E. Family connections: a program for relatives of persons with borderline personality disorder. Fam Process. 2005 Jun;44(2):217-25. doi: 10.1111/j.1545-5300.2005.00055.x. PMID 16013747
- [Background] Hoffman PD, Buteau E, Hooley JM, Fruzzetti AE, Bruce ML. Family members' knowledge about borderline personality disorder: correspondence with their levels of depression, burden, distress, and expressed emotion. Fam Process. 2003 Winter;42(4):469-78. doi: 10.1111/j.1545-5300.2003.00469.x. PMID 14979218
- [Background] Hoffman PD, Fruzzetti AE, Swenson CR. Dialectical behavior therapy--family skills training. Fam Process. 1999 Winter;38(4):399-414. doi: 10.1111/j.1545-5300.1999.00399.x. PMID 10668619
- [Background] Flynn D, Kells M, Joyce M, Corcoran P, Herley S, Suarez C, Cotter P, Hurley J, Weihrauch M, Groeger J. Family Connections versus optimised treatment-as-usual for family members of individuals with borderline personality disorder: non-randomised controlled study. Borderline Personal Disord Emot Dysregul. 2017 Aug 30;4:18. doi: 10.1186/s40479-017-0069-1. eCollection 2017. PMID 28861273
- [Background] Rajalin M, Wickholm-Pethrus L, Hursti T, Jokinen J. Dialectical behavior therapy-based skills training for family members of suicide attempters. Arch Suicide Res. 2009;13(3):257-63. doi: 10.1080/13811110903044401. PMID 19590999
- [Background] Liljedahl SI, Kleindienst N, Wangby-Lundh M, Lundh LG, Daukantaite D, Fruzzetti AE, Westling S. Family Connections in different settings and intensities for underserved and geographically isolated families: a non-randomised comparison study. Borderline Personal Disord Emot Dysregul. 2019 Aug 26;6:14. doi: 10.1186/s40479-019-0111-6. eCollection 2019. PMID 31463066
- [Derived] Marco JH, Fonseca S, Fernandez-Felipe I, Garcia-Palacios A, Banos R, Perez S, Garcia-Alandete J, Guillen V. Family connections vs treatment at usual optimized in the treatment of relatives of people with suicidal behavior disorder: study protocol of a randomized control trial. BMC Psychiatry. 2022 May 15;22(1):335. doi: 10.1186/s12888-022-03965-5. PMID 35570289